CLINICAL TRIAL: NCT01688843
Title: INGEVITY(TM) Active Fixation and Passive Fixation Pace/ Sense Lead Clinical Study
Brief Title: Safety and Performance Study of the INGEVITY Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSC-CDM00048360
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2017-11-17 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Bradycardia; Sinus Node Dysfunction
Keywords: bradycardia; sinus node dysfunction
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INGEVITY lead (Experimental): INGEVITY lead implant
  Interventions: Device: INGEVITY lead

INTERVENTIONS:
Device: INGEVITY lead

SUMMARY:
The objective of this study is to gather data to establish the safety, performance and effectiveness of the INGEVITY pace/ sense leads.

DETAILED DESCRIPTION:
The objective of this study is to gather data to establish the safety, performance and effectiveness of the INGEVITY pace/ sense leads

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and capable of providing informed consent
* Subject has a Class I or II indication for implantation of a single(VVI (R) only) or dual chamber pacemaker or a CRT-P system according to the ACC/AHA/HRS, or ESC guidelines
* Subject is willing and capable of participating in all testing/ visits associated with this clinical study at an approved clinical study center and at the intervals defined by this protocol
* Subject is age 18 or above, or of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Subject has or has had any pacing or ICD system implants
* Subject has a sensitivity to dexamethasone acetate (DXA)
* Subject has a mechanical tricuspid heart valve
* Subject is enrolled in any other concurrent study, with the exception of local mandatory governmental registries and observational studies/registries
* Subjects with documented permanent or persistent AF where the physician intends to implant dual chamber pulse generator (single chamber VVIR pulse generators in these subjects is acceptable)
* Subject is currently on the active heart transplant list
* Subject has documented life expectancy of less than 12 months
* Women of childbearing potential who are or might be pregnant at the time of study enrollment or INGEVITY Lead implant
* Subjects currently requiring dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1060 (Actual)
Dates: Start 2012-10; Primary Completion 2015-01 (Actual); Study Completion 2019-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Love, MD, Principal Investigator — Johns Hopkins University
Locations (78):
- United States (44):
  - Mercy Gilbert Medical Center, Gilbert, Arizona
  - Cardiovascular Consultants, LTD, Glendale, Arizona
  - Pima Heart Physicians, PC, Tucson, Arizona
  - Sharp Grossmont Hospital, La Mesa, California
  - Orange County Heart Institute, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Sharp Memorial Hospital, San Diego, California
  - Danbury Hospital, Danbury, Connecticut
  - Cardiology Associates of Fairfield County, Trumbull, Connecticut
  - West Florida Cardiology Network, LLC, Largo, Florida
  - University Community Hospital, Tampa, Florida
  - Wellstar Research Institute, Marietta, Georgia
  - St. Vincent's Hospital, Indianapolis, Indiana
  - Indiana University Health La Porte Hospital, La Porte, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Southern Kentucky Heart Institute, Bowling Green, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan CardioVascular Institute, Saginaw, Michigan
  - HealthEast St. Joseph's Hospital, Saint Paul, Minnesota
  - Cardiovascular Associates of the Delaware Valley, Sewell, New Jersey
  - New York Methodist Hospital, Brooklyn, New York
  - Rochester General Hospital, Rochester, New York
  - Staten Island University Hospital, Staten Island, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - Lindner Center for Research and Education at Christ Hosp, Cincinnati, Ohio
  - University Hospital, Inc., Cincinnati, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Coastal Cardiology, Charleston, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - South Austin Hospital, Austin, Texas
  - Heart Hospital of Austin, Austin, Texas
  - North Texas Heart Center, Dallas, Texas
  - Plaza Medical Center of Fort Worth, Fort Worth, Texas
  - Trinity Mother Frances Health System, Tyler, Texas
  - University of Utah Hospital and Clinics, Salt Lake City, Utah
  - Bon Secours Heart & Vascular Institute, Richmond, Virginia
  - PeaceHealth St. Joseph Medical Center, Bellingham, Washington
  - Monongalia General Hospital, Morgantown, West Virginia
  - Wheeling Hospital Inc., Wheeling, West Virginia
  - Wheaton Franciscan Healthcare, Glendale, Wisconsin
  - St. Mary's Madison, Madison, Wisconsin
- Australia (2):
  - St. Andrew's War Memorial Hospital, Brisbane, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
- Austria (3):
  - Medizinische Univ.-Kliniken Graz, Graz
  - AKH Linz, Linz
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge Campus, Kortrijk
- Canada (3):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - Hamilton General Hospital, Hamilton, Ontario
  - Hopital Hotel Dieu du Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
- Denmark (2):
  - Skejby Sygehus, Aarhus
  - Roskilde University Hospital, Roskilde
- France (2):
  - CHU La Timone Hospital, Marseille
  - NCN Nouvelles Cliniques Nantaises, Nantes
- Germany (4):
  - Kardiologische Gemeinschaftspraxis Kaltofen Schubert Gerner, Chemnitz
  - Uniklinik Köln, Cologne
  - Universitätsklinikum Erlangen, Erlangen
  - Otto-von-Guericke-Universitaet Magdeburg, Magdeburg
- Prince of Wales Hospital, Shatin, Hong Kong
- Azienda Ospedaliera Universitaria Integrata di Verona, Verona, Italy
- Malaysia (2):
  - Institut Jantung Negara, Kuala Lumpur
  - University of Malaya Medical Centre, Kuala Lumpur
- Portugal (2):
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto
  - Hospital de Santarem, Santarém
- Spain (4):
  - Hospital Clinico Y Provincial, Barcelona
  - Hospital Universitario Nuestra Senora de Candelaria, Santa Cruz de Tenerife
  - Hospital Doctor Peset, Valencia
  - Clinico de Valladolid, Valladolid
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
- Chiang Mai Heart Center Medical School Hospital, Chiang Mai, Thailand
- United Kingdom (3):
  - Basildon and Thurrock University Hospitals NHS, Basildon, Essex
  - Belfast City Hospital, Belfast
  - Wrexham Maelor Hospital, Wrexham

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Leads
Groups:
- INGEVITY Study Participants: Each participant was allowed to have up to 2 INGEVITY leads contribute to endpoint analyses -- one per chamber (right atrium and right ventricle). Final lead implanted or attempted during initial procedure per chamber was used for analysis.
Period: Overall Study
Arm/Group | INGEVITY Study Participants
Started | 1060; 1599 Leads
Completed | 1060; 1599 Leads
Not Completed | 0; 0 Leads

BASELINE CHARACTERISTICS:
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 1060
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 478
  Male | 582
Region of Enrollment [Number; unit: participants]
  Hong Kong | 11
  United States | 603
  United Kingdom | 39
  Malaysia | 25
  Thailand | 10
  Portugal | 32
  Spain | 88
  Canada | 20
  Austria | 45
  Sweden | 16
  Belgium | 22
  Denmark | 26
  Italy | 21
  Australia | 8
  France | 57
  Germany | 37

OUTCOME MEASURES:

1. Primary Outcome: Safety 1 - Percentage of Leads Free From Complication (0 - 3 Months)
Description: Lead-related complication-free rate from lead implant through the three month follow-up, based on complications that are related to the INGEVITY Lead. The performance goal based on similar leads was set in collaboration with FDA at 91.4%
Time Frame: Lead implant through 3 month follow up
Population: Final lead implanted or attempted during initial procedure per chamber was used for analysis. Analysis leads were from participants who met inclusion/exclusion criteria and were implanted or attempted with INGEVITY lead(s). Of the 1060 enrolled participants, 24 did not meet these criteria and were excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of leads complication-free
Units Other Than Participants: Implant/Attempted Leads
Groups:
- INGEVITY Lead: Implanted/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 1036
Number analyzed (Implant/Attempted Leads) | 1599
percentage of leads complication-free | 98.4 [97.7 to NA] — One-sided confidence interval

2. Primary Outcome: Safety 2 - Percentage of Leads Free From Complication (3 - 24 Months)
Description: Lead-related complication-free rate from three months post-implant through twelve months post implant, based on complications that are related to the INGEVITY Lead. The performance goal based on similar leads was set in collaboration with FDA at 94%.
Time Frame: 3 months through 12 months post implant
Population: Leads still in service and implanted in actively followed participants at 92 days were included in analysis.
Measure: Number (95% Confidence Interval); unit: percentage of leads complication-free
Units Other Than Participants: Implant/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 1009
Number analyzed (Implant/Attempted Leads) | 1545
percentage of leads complication-free | 99.7 [99.4 to NA] — One-sided confidence interval

3. Primary Outcome: Safety 3 - Hazard Rate of Lead-Related Complications
Description: Hazard rate of lead-related complications over time. This endpoint will use the Weibull distribution to estimate the hazard over time by evaluating the Weibull shape parameter. A Weibull shape greater than one (>1), equal to one (=1) and less than one (<1) indicates accelerating, constant, and decelerating hazard of lead-related complications over time, respectively. This endpoint requires the Weibull shape estimate to be less than 1.
Time Frame: Implant through 12 months (including available data beyond 12 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: hazard rate of lead-related complication
Units Other Than Participants: Leads Implanted/Attempted
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 1036
Number analyzed (Leads Implanted/Attempted) | 1599
hazard rate of lead-related complication | 0.23 [NA to 0.3] — One-sided confidence interval

4. Primary Outcome: Effectiveness 1
Description: The bipolar pacing threshold at 0.5 ms at three months post-implant < 1.5 V
Time Frame: Lead implant through 3 month follow up
Measure: Mean (95% Confidence Interval); unit: volts
Units Other Than Participants: Implant/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 982
Number analyzed (Implant/Attempted Leads) | 1482
volts | 0.67 [0.65 to 0.69]

5. Primary Outcome: Effectiveness 2(Right Atrium)
Description: P-wave sensed amplitude at three months post-implant > 1.5 mV
Time Frame: Lead implant through 3 month follow up
Measure: Mean (95% Confidence Interval); unit: mV
Units Other Than Participants: Implant/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 521
Number analyzed (Implant/Attempted Leads) | 521
mV | 4.8 [4.6 to NA] — One-sided confidence interval

6. Primary Outcome: Effectiveness 2(Right Ventricle)
Description: R-wave sensed amplitude at three months post-implant > 5 mV
Time Frame: Lead implant through 3 month follow up
Measure: Mean (95% Confidence Interval); unit: mV
Units Other Than Participants: Implant/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 914
Number analyzed (Implant/Attempted Leads) | 914
mV | 16.5 [16.2 to NA] — One-sided confidence interval

7. Primary Outcome: Effectiveness 3
Description: Clinically acceptable pacing impedance between 300 Ω and 1300 Ω
Time Frame: Lead implant through 3 month follow up
Measure: Mean (95% Confidence Interval); unit: Ω
Units Other Than Participants: Implant/Attempted Leads
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 995
Number analyzed (Implant/Attempted Leads) | 1526
Ω | 773 [766 to 779]

8. Other Pre Specified Outcome: Ancillary Safety
Description: Lead-related complication-free rate
Time Frame: From 3 to 60 months post-implant
Population: Leads eligible for endpoint analyses
Measure: Number (95% Confidence Interval); unit: percentage of leads complication-free
Units Other Than Participants: Leads
Groups:
- INGEVITY Lead: INGEVITY lead implant
  INGEVITY lead
Arm/Group | INGEVITY Lead
Number analyzed (Participants) | 1038
Number analyzed (Leads) | 1599
percentage of leads complication-free | 99.1 [98.6 to 100]

ADVERSE EVENTS:
Time Frame: Entire follow-up (median participant follow-up = 30.9 months)
Description: All-cause mortality evaluated in all enrolled participants (N = 1060). Adverse events evaluated in participants implanted or attempted with at least one INGEVITY lead (N = 1041). Individual adverse event categories evaluated in participants at risk for that event category (e.g., Pulse generator events evaluated in participants with a pulse generator).
Arm/Group | INGEVITY Study Participants
All-Cause Mortality (participants affected / at risk) | 93/1060
Serious Adverse Events (participants affected / at risk) | 532/1041
Other Adverse Events (participants affected / at risk) | 621/1041
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | INGEVITY Study Participants (N=1041)
Pulse Generator (Product Issues) | 9 (10) — Includes: Oversensing - Defibrillation Rate response inappropriate Inappropriate AV delay Pacemaker-mediated tachycardia (PMT) Erosion Infection (> 30 days post-implant) Migration
Right Atrial (RA) Lead - INGEVITY Related (Product Issues) | 10/564 (10) — 564 patients were attempted/implanted with a INGEVITY RA lead, therefore that is the number at risk for an adverse event
RA Lead - Other (Non-INGEVITY Lead) (Product Issues) | 12/858 (12) — 858 patients were attempted/implanted with an OTHER (non-INGEVITY) RA lead, therefore that is the number at risk for an adverse event
Right Ventricular (RV) Lead - INGEVITY-related (Product Issues) | 15 (20) — Includes: Unable to capture - RV - INGEVITY-related Elevated threshold - RV - INGEVITY-related Extracardiac stimulation - RV - INGEVITY-related Conductor coil fracture - RV - INGEVITY-related Dislodgment - RV - INGEVITY-related
RV Lead - Other (Non-INGEVITY Lead) (Product Issues) | 1 (1) — Includes: Other - RV Lead - Other
Left-Ventricular (LV) Lead (Product Issues) | 2 (2) — Includes: Elevated threshold - LV Extracardiac stimulation - LV Dislodgment - LV
Procedure (Surgical and medical procedures) | 26 (26)
Cardiovascular - Heart Failure (Cardiac disorders) | 101 (163)
Cardiovascular - Non-Heart Failure (Cardiac disorders) | 241 (326)
Other (General disorders) | 49 (54)
Unclassified (Investigations) | 8 (8)
Non-cardiovascular (General disorders) | 357 (705)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | INGEVITY Study Participants (N=1041)
Pulse Generator (Product Issues) | 32 (37)
RA Lead - INGEVITY-related (Product Issues) | 16/564 (17) — 564 patients were attempted/implanted with an INGEVITY RA lead, therefore that is the number at risk for an adverse event
RA Lead - Other (Product Issues) | 4/858 (4) — 858 patients were attempted/implanted with an OTHER (non-INGEVITY) RA lead, therefore that is the number at risk for an adverse event
RV Lead - INGEVITY-related (Product Issues) | 11 (11)
LV Lead (Product Issues) | 6/47 (7) — 47 patients were attempted/implanted with any LV lead, therefore that is the number at risk for an adverse event
Procedure (Surgical and medical procedures) | 58 (66)
Cardiovascular - HF (Cardiac disorders) | 61 (74)
Cardiovascular - Non-HF (Cardiac disorders) | 412 (720)
Other (General disorders) | 89 (103)
Unclassified (General disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No